CLINICAL TRIAL: NCT03361917
Title: Prospective Randomized Controlled Trial of High-Definition White-light Colonoscopy Versus High-Definition White-light Colonoscopy With Endocuff Vision for Endpoints of Procedural Times
Brief Title: Standard Colonoscopy Versus Colonoscopy With Endocuff Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Distinguished Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1709336500; NCT03398447 (obsolete NCT alias)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2019-05-22 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Polyp; Colorectal Adenoma; Colon Cancer
Keywords: Colonoscopy screening; Colonscopy procedure
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Arm (Standard Colonscopy) (No Intervention): Standard colonoscopy with no device attachments
- Endocuff Vision (Experimental): Colonoscopy with Endocuff Vision attached to distal end of scope
  Interventions: Device: Endocuff Vision

INTERVENTIONS:
Device: Endocuff Vision — Subjects that are randomized to undergo their colonoscopy procedure with the Endocuff Vision device will have the device placed on the colonoscope that will be used during their procedure.
  Arms: Endocuff Vision

SUMMARY:
This study seeks to compare colonoscopy results between a standard method and one using a distal scope attachment (Endocuff Vision).

DETAILED DESCRIPTION:
For this study, subjects will be randomized into one of two groups (those who receive a standard colonoscopy and those who receive a colonoscopy with an Endocuff Vision attachment). Results will then be compared between the two; these include insertion time (time it takes to reach the cecum of the large intestine), inspection time (time spent examining the large intestine), the total time per each polypectomy (removal of polyps in the colon), and the total procedure time of the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for a screening or surveillance colonoscopy
* Subject is aged 40 years or older
* Subject has the ability to provide informed consent

Exclusion Criteria:

* Prior history of colon cancer
* History of inflammatory bowel disease
* Prior surgical resection of any part of the colon
* Use of antiplatelet agents or anticoagulants that precludes the removal of polyps during the procedure
* History of polyposis syndrome or HNPCC
* Family history of colon cancer in a first-degree relative < 60 years or two first degree relatives with colorectal cancer
* Inability to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data can be shared in the future upon request.

REFERENCES:
- [Background] Tsiamoulos ZP, Misra R, Rameshshanker R, Elliott TR, Beintaris I, Thomas-Gibson S, Haycock A, Suzuki N, Rees C, Saunders BP. Impact of a new distal attachment on colonoscopy performance in an academic screening center. Gastrointest Endosc. 2018 Jan;87(1):280-287. doi: 10.1016/j.gie.2017.04.001. Epub 2017 Apr 13. PMID 28412271
- [Derived] Rex DK, Slaven JE, Garcia J, Lahr R, Searight M, Gross SA. Endocuff Vision Reduces Inspection Time Without Decreasing Lesion Detection: A Clinical Randomized Trial. Clin Gastroenterol Hepatol. 2020 Jan;18(1):158-162.e1. doi: 10.1016/j.cgh.2019.01.015. Epub 2019 Jan 17. PMID 30659990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm (Standard Colonscopy) | Endocuff Vision
Started | 99 | 101
Completed | 99 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy) | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (8.9) | 61.7 (9.9) | 62.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 57 | 101
  Male | 57 | 42 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 92 | 179
  Other | 14 | 7 | 21
Region of Enrollment [Number; unit: participants]
  United States | 101 | 99 | 200
Gastroenterology fellows assisting in insertion [Count of Participants; unit: Participants] | 17 | 15 | 32
Procedure Indication [Count of Participants; unit: Participants]
  Screening | 45 | 52 | 97
  Surveillance | 56 | 47 | 103

OUTCOME MEASURES:

1. Primary Outcome: Inspection Time Comparisons for Each Method (Standard vs. Endocuff Vision)
Description: Inspection time is time spent actually examining the colon. This was measured with a stopwatch and calculated by subtracting washing, suctioning, polypectomy and biopsy times from total withdrawal time. It was measured during colonoscopy by a study assistant using a stopwatch.
Time Frame: During the withdrawal portion of the colonoscopy procedure
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy)
Number analyzed (Participants) | 101 | 99
Minutes | 6.49 (.10) | 8.42 (0.12)

2. Secondary Outcome: Insertion Time Comparisons for Each Method (Standard vs. Endocuff Vision)
Description: Insertion time is the time it takes from the colonoscope first being inserted to when the furthest section of the colon (which is called the cecum) is reached.
Time Frame: During the insertion portion of the colonoscopy procedure
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy)
Number analyzed (Participants) | 101 | 99
Minutes | 4.05 (0.16) | 4.42 (0.19)

3. Secondary Outcome: Total Procedure Time Comparisons for Each Method (Standard vs. Endocuff Vision)
Description: Total procedure time is the time from the initial insertion through the complete withdrawal of the scope
Time Frame: During the colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy)
Number analyzed (Participants) | 101 | 99
Minutes | 21.01 (6.8) | 21.24 (7.8)

4. Secondary Outcome: Detection Rates
Description: The percentage of participants with at least one of the indicated polyp types found during standard colonoscopy compared to colonoscopy with Endocuff Vision.
Time Frame: During the colonoscopy procedure
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy)
Number analyzed (Participants) | 101 | 99
Percentage of Participants
  Adenomas | 61.4 [51.6 to 70.3] | 52.5 [42.8 to 62.1]
  Sessile serrated polyps | 19.8 [13.2 to 28.6] | 11.1 [6.3 to 18.8]

5. Secondary Outcome: Polyps Per Colonoscopy
Description: Number of adenomas or sessile serrated polyps found per colonoscopy of Standard colonoscopy compared to Colonoscopy with Endocuff Vision.
Time Frame: During the colonoscopy procedure
Measure: Mean (Standard Error); unit: Polyps per colonoscopy
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy)
Number analyzed (Participants) | 101 | 99
Polyps per colonoscopy
  Adenomas | 1.43 (1.79) | 1.07 (1.62)
  Sessile serrated polyps | 0.27 (0.63) | 0.21 (0.70)

6. Secondary Outcome: Boston Bowel Preparation Score
Description: Boston Bowel Preparation Score for patients receiving standard colonoscopy compared to colonoscopy with endocuff vision.
  The total score for the Boston Bowel Preparation Scale ranges from 0 to 9, with higher score indicating a better bowel preparation quality.
  The quality of the bowel preparation is assessed by the attending gastroenterologist.
Time Frame: During the withdrawal portion of the colonoscopy procedure after cleaning of the colon
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Endocuff Vision | Control Arm (Standard Colonscopy)
Number analyzed (Participants) | 101 | 99
Scores on a scale | 9 [3 to 9] | 9 [3 to 9]

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Control Arm (Standard Colonscopy) | Endocuff Vision
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/101
Other Adverse Events (participants affected / at risk) | 0/99 | 0/101

LIMITATIONS AND CAVEATS:
Examiners were not blinded to the device used. Only 2 examiners with experience with the device participated in the study so generalizability of the results is unknown.

Data was not collected on other potential confounders like smoking or BMI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03361917/Prot_SAP_000.pdf